CLINICAL TRIAL: NCT06754254
Title: Performance of Blood Biomarkers in Different Circulation Sites on Detecting Alzheimer's Pathologies - the Delta Study
Brief Title: Blood Biomarkers from Internal Jugular Vein for the Diagnosis of Alzheimer's Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yan-Jiang Wang, Prof., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: IJV-AD-24
Record Dates: First submitted 2024-07-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and cerebrospinal fluid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Aβ PET (+)
  Interventions: Diagnostic Test: blood biomarkers from the internal jugular vein
- Aβ PET (-)
  Interventions: Diagnostic Test: blood biomarkers from the internal jugular vein

INTERVENTIONS:
Diagnostic Test: blood biomarkers from the internal jugular vein — blood biomarkers (Aβ42/40, p-tau217, p-tau181, NFL, GFAP, etc.) from the internal jugular vein

SUMMARY:
The goal of this observational study is to explore the diagnostic performance of blood biomarkers from the internal jugular vein for the diagnosis of Alzheimer's disease (AD) in patients with cognitive symptoms or concerns. The main question it aims to answer is:

Whether blood biomarkers from the internal jugular vein outperform those from the median cubital vein which is the routine site for venous blood collection?

ELIGIBILITY:
Inclusion Criteria:

1. age: 40-90 years old (including 40 and 90 years);
2. patients with cognitive complaints or concerns;
3. Willing and able to comply with all aspect of the protocol and provide written informed consent. If a subject lacks capacity to consent in the investigator's opinion, the subject's assent should be obtained, if required in accordance with local laws, regulations and customs, plus the written informed consent of a legal representative should be obtained (capacity to consent and definition of legal representative should be determined in accordance with applicable local laws and regulations).

Exclusion Criteria:

1. Severe medical conditions which are not stably and could affect the subject's safety;
2. Presence of contraindications for PET examination, cerebrospinal fluid or blood collection;
3. Unwilling and refuse to participate in this study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cognitive symptoms or concerns were consectively recruited from memory clinics.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | 5 years from the enrollment of the first participant
  area under the ROC curve, accuracy, sensitivity, specificity, positive predictive value, negative predictive value

SECONDARY OUTCOMES:
Correlation with CSF biomarkers | 5 years from the enrollment of the first participant
  Correlations of blood biomarkers (Aβ42, Aβ40, Aβ42/40 ratio, p-tau217, p-tau181, p-tau217/Aβ42 ratio, p-tau181/Aβ42 ratio, NFL, GFAP, etc.) with CSF biomarkers (Aβ42，Aβ40， Aβ42/40 ratio, p-tau181，p-tau181/Aβ42 ratio, GFAP，NFL, etc.).
Correlation with brain Aβ burden | 5 years from the enrollment of the first participant
  Correlations of blood biomarkers (Aβ42, Aβ40, Aβ42/40 ratio, p-tau217, p-tau181, p-tau217/Aβ42 ratio, p-tau181/Aβ42 ratio, NFL, GFAP, etc.) with brain Aβ burden measured by Aβ PET.
Correlation with brain Tau burden | 5 years from the enrollment of the first participant
  Correlations of blood biomarkers (Aβ42, Aβ40, Aβ42/40 ratio, p-tau217, p-tau181, p-tau217/Aβ42 ratio, p-tau181/Aβ42 ratio, NFL, GFAP, etc.) with brain tau burden measured by Tau PET.
Effects of comorbidities on blood biomarkers and diagnostic performance | 5 years from the enrollment of the first participant
  Associations (beta value) of comorbidites (hypertension, diabetes, history of stroke or myocardial infarction, hepatic or renal insufficiency, etc.) with the levels of blood biomarkers (Aβ42, Aβ40, Aβ42/40 ratio, p-tau217, p-tau181, p-tau217/Aβ42 ratio, p-tau181/Aβ42 ratio, NFL, GFAP, etc.) and their diagnostic performance (area under the curve, accuracy, sensitivity, specificity, positive predictive value, negative predictive value).

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No